CLINICAL TRIAL: NCT00629889
Title: Levetiracetam and Pregabalin for Monotherapy in Patients With Brain Tumors and Seizures. A Phase II Randomized Study.
Brief Title: Levetiracetam or Pregabalin in Treating Seizures in Patients Undergoing Chemotherapy and/or Radiation Therapy For Primary Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr Andrea Rossetti (Other)
Responsible Party: Sponsor-Investigator, Dr Andrea Rossetti, Médecin associé, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000586523; CHUV-Neurology-CePO-LEV-PGB; EU-20807
Record Dates: First submitted 2008-03-05; First posted 2008-03-06 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Brain and Central Nervous System Tumors; Seizure
Keywords: seizure; adult anaplastic astrocytoma; adult diffuse astrocytoma; adult pineal gland astrocytoma; adult glioblastoma; adult gliosarcoma; adult giant cell glioblastoma; adult brain stem glioma; adult ependymoblastoma; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult ependymoma; adult anaplastic ependymoma; adult anaplastic meningioma; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult pineoblastoma; adult pineocytoma; adult mixed glioma; adult papillary meningioma; recurrent adult brain tumor; adult grade II meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Seizures; Astrocytoma; Glioblastoma; Gliosarcoma; Neuroectodermal Tumors, Primitive; Medulloblastoma; Ependymoma; Meningioma; Oligodendroglioma; Pinealoma; Glioma; Brain Neoplasms | interventions — Levetiracetam; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Active Comparator): Patients assigned to Levetiracetam are treated with the initial dose of 2 x 250mg per day up to one year
  Interventions: Drug: pregabalin
- Pregabalin (Active Comparator): Patients assigned to Pregabalin are treated with the initial dose of 2 x 75mg per day up to one year
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam — After inclusion, patients receive Levetiracetam 2x250mg per day. The medication may be increased, in intervals of 500mg of Levetiracetam of at least 24h up to maximally: Levetiracetam 2x1500mg.
  Patients might be treated up to one year within the study. If well tolerated, treatment might continue after end of study.
  Arms: Pregabalin
Drug: pregabalin — After inclusion, patients receive Pregabalin 2x75mg per day. The medication may be increased, in intervals of 150mg of Pregabalin of at least 24h up to maximally: Pregabalin 2x300mg.
  Patients might be treated up to one year within the study. If well tolerated, treatment might continue after end of study.
  Arms: Levetiracetam

SUMMARY:
RATIONALE: Levetiracetam and pregabalin are drugs that treat seizures. It is not yet known which drug is more effective in treating seizures caused by primary brain tumors.

PURPOSE: This randomized phase II trial is studying the side effects and how well levetiracetam or pregabalin work in treating seizures in patients undergoing chemotherapy and/or radiation therapy for primary brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the safety and efficacy of antiepileptic drug monotherapy comprising levetiracetam or pregabalin in treating seizures in patients undergoing chemotherapy and/or radiotherapy for primary brain tumors.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive levetiracetam.
* Arm II: Patients receive pregabalin. Patients are followed at 2 weeks, 2 months, 6 months, and then at 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary brain tumor

  * WHO grade II-IV disease
* Undergoing chemotherapy and/or radiotherapy
* No brain tumor without the potential need for chemotherapy (e.g., meningioma without anaplastic features)
* Has had at least one seizure provoked by the brain tumor, justifying introduction of antiepileptic drug (AED) treatment

  * No status epilepticus

PATIENT CHARACTERISTICS:

* Modified Rankin score < 4 at study enrollment
* Life expectancy ≥ 4 weeks
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known intolerance to the study drugs
* No pre-existing psychosis and/or current suicidality

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent IV AEDs other than benzodiazepines
* Other concurrent AEDs, except phenobarbital, allowed provided they are discontinued within 2 weeks after study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-02; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Survival without occurrence of status epilepticus, 2 seizures with consciousness impairment, need to add a second antiepileptic drug (AED) (except transitory benzodiazepine), and need to discontinue study drug for lack of efficacy or adverse events | baseline to visit at 12 months

SECONDARY OUTCOMES:
Adverse events | baseline to visit at 12 months
Anxiety | baseline to visit at 12 months
Need to add a second AED | baseline to visit at 12 months
Study drug discontinuation | baseline to visit at 12 months
Occurrence of consciousness-impairing seizures or status epilepticus | baseline to visit at 12 months
Mortality | baseline to visit at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea O. Rossetti, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (2):
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - USZ, Zurich